CLINICAL TRIAL: NCT01511133
Title: Blinded Retrospective Laboratory Evaluations to Assess the Serologic Response to Porcine Circovirus Type 1 (PCV-1) and PCV-1 DNA in the Stool of Infants Aged 6 to 12 Weeks Following Administration of GlaxoSmithKline (GSK) Biologicals' Oral Live Attenuated Human Rotavirus Vaccine (444563)
Brief Title: Serological Response to Porcine Circovirus Type 1 (PCV-1) and PCV-1 DNA in Stools of Infants Following Administration of Rotarix™
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114444; 444563/022 (Other: GSK); 444563/033 (Other: GSK); 103477 (Other: GSK); 104480 (Other: GSK)
Record Dates: First submitted 2011-12-01; First posted 2012-01-18 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Rotavirus Infection; Evidence of PCV-1 Replication and/or Immune Response to the PCV-1 in HRV Vaccinated Infants
Keywords: Laboratory evaluations; infants; Porcine circovirus type 1 (PCV-1); serologic response; human rotavirus (HRV) vaccine
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum and stool samples

GROUPS / COHORTS (2):
- HRV Group: Subjects received two or three doses of HRV in previous studies.
  Interventions: Procedure: Stool sample; Procedure: Serum sample
- Placebo Group: Subjects received two or three doses of placebo in previous studies.
  Interventions: Procedure: Stool sample; Procedure: Serum sample

INTERVENTIONS:
Procedure: Stool sample — Stool samples collected at pre-determined time points in previous studies will be analysed to detect the presence of PCV-1 DNA and pattern of detection.
Procedure: Serum sample — Serum samples collected at pre and post vaccination time points in previous studies will be assessed for Anti-PCV-1 antibody.

SUMMARY:
This study aims to test the clinical samples (stool and serum) previously collected during clinical development of HRV vaccine, to identify if there is any evidence of PCV-1 replication and/or immune response to the PCV-1 in vaccinated infants.

DETAILED DESCRIPTION:
Serum and stool samples collected from 4 clinical trials previously conducted for HRV vaccine (Rotarix™) are used in this study.

ELIGIBILITY:
Inclusion criteria:

* Subjects enrolled previously in randomized, double-blind and placebo-controlled studies 444563/022 (NCT00263666), 444563/033 (NCT00757770), 103477 (NCT00169455), and 104480 (NCT00137930);
* Infants aged 6 to 12 weeks at Dose 1 vaccinated with either HRV vaccine or placebo;
* Infants for whom sufficient residual volume of the stool samples at predetermined time points is available;
* Infants for whom sufficient residual volume of the pre and post vaccination blood samples is available.

Exclusion criteria:

- Not applicable

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants aged 6 to 12 weeks from 4 previously conducted clinical trials, who received 2 or 3 doses of either Rotarix™ or Placebo
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Presence of PCV-1 DNA and pattern of detection in the stool samples collected | At pre-defined time points after vaccination (3-7 time points up to day 45 after vaccination)
Presence of serum anti-PCV-1 antibody | At pre and post vaccination time points (At Day 0 and 2 Months after last dose vaccination)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Han HH, Karkada N, Jayadeva G, Dubin G. Serologic response to porcine circovirus type 1 (PCV1) in infants vaccinated with the human rotavirus vaccine, Rotarix: A retrospective laboratory analysis. Hum Vaccin Immunother. 2017 Jan 2;13(1):237-244. doi: 10.1080/21645515.2016.1231262. PMID 27657348